CLINICAL TRIAL: NCT03072732
Title: Measuring Thoracic Impedance in Hemodialysis Patients With the µ-Cor System A Pre-Market Validation Study (MaTcH)
Brief Title: Measuring Thoracic Impedance in Hemodialysis Patients With the u-Cor Monitoring System
Acronym: MaTcH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-KM-004
Record Dates: First submitted 2017-03-01; First posted 2017-03-07 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Fluid Retention Tissue
Keywords: Heart Failure; Hemodialysis
MeSH Terms: conditions — Edema; Heart Failure

STUDY DESIGN:
Intervention Model Description: 2-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- study arm 1 - below left axilla (Other): 20 patients undergoing hemodialysis, with at least 10 of these patients having congestive heart failure, will have the u-Cor system placed below left axilla and the ZOE Fluid Status Monitor
  Interventions: Device: u-Cor System; Device: ZOE Fluid Status Monitor
- study arm 2-upper left pectoral area (Other): 20 patients undergoing hemodialysis, with at least 10 of these patients having congestive heart failure, will have the u-Cor system placed on the upper left pectoral area and the ZOE Fluid Status Monitor
  Interventions: Device: u-Cor System; Device: ZOE Fluid Status Monitor

INTERVENTIONS:
Device: u-Cor System — Monitoring System
  Other Names: u-Cor V3.0 System
Device: ZOE Fluid Status Monitor — Monitoring System

SUMMARY:
The purpose of this study is to measure the fluid changes in the body using a device called the µ-Cor System, an investigational device. The µ-Cor System will record the fluid changes in the body, as well as ECG (electrocardiogram or an electrical tracing of your heart rhythm) heart rate, breathing rate, posture and activity at regular intervals.

The information collected by the µ-Cor System will then be compared to the actual fluid removed through dialysis and to the information collected by an FDA (Food and Drug Administration) cleared device called ZOE (NonInvasive Medical Technologies), a monitor which also measures the fluid changes in the body.

The objectives of this study are to document any differences in measurement of thoracic impedance obtained from the µ-Cor System and the ZOE system. Thoracic impedance is a measure of the electrical activity in the chest that varies with changes in body size and composition, fluid volume, breathing status and other variables.

Measurements of the amount of fluid removed during dialysis will also be compared between the µ-Cor System, the ZOE system and the actual fluid removed.

The ability of the µ-Cor System to measure thoracic impedance will be tested by placing the device randomly at one of two locations:

* Study Arm 1: side location- below left axilla
* Study Arm 2: front location - upper left pectoral area

Both the µ-Cor System and the ZOE System will be worn simultaneously during one dialysis session. The ZOE system device is placed on the chest- 2 points: 1 at the base of your neck and 1 in your mid chest.

DETAILED DESCRIPTION:
The µ-Cor System is intended to record, store, transmit, and display the following physiological data to medical professionals: thoracic impedance, ECG, heart rate, respiration rate, activity and posture.

The µ-Cor System is indicated for patients who are 21 years of age or older who:

* have fluid-management problems,
* are taking diuretic medication,
* are living with heart failure,
* are living with end-stage renal disease,
* are recovering from a coronary artery disease-related event, and/or
* are suffering from recurrent dehydration.

Objectives:

* This clinical trial is intended to provide evidence of substantial equivalence between the µ-Cor System and the ZOE System in the ability to measure thoracic impedance, by comparing the correlation between µ Cor measurement and ultrafiltration volume (UFV) as compared with the correlation between ZOE measurement and UFV. The actual UFV changes will be used to arbitrate any differences.
* The ability of the µ-Cor System to measure thoracic impedance will be demonstrated at 2 body locations: side location (below left axilla, Study Arm 1), and front location (upper left pectoral area, Study Arm 2).

Subject population:

Forty patients undergoing hemodialysis (n = 40) in 2 study arms with at least 50% enrollment of patients diagnosed with congestive heart failure (CHF) in each arm:

* Study Arm 1: 20 patients undergoing hemodialysis, with at least 10 of these patients having CHF, will have the µ-Cor device placed on the side location
* Study Arm 2: 20 patients undergoing hemodialysis, with at least 10 of these patients having CHF, will have the µ-Cor device placed on the front location

Patients will wear the µ-Cor device and will be connected to the ZOE monitor during one hemodialysis session in the clinic. Patients will be randomly allocated to Study Arm 1 or Study Arm 2, with randomization stratified by CHF status (CHF or non-CHF). During the hemodialysis session, the patient will wear 1 µ-Cor device and will be connected simultaneously to 1 ZOE monitor (via 2 ZOE electrodes) for comparative measurements and UFV correlation, from at least 15 minutes before the start of dialysis to at least 15 minutes after the end of the dialysis session. The µ-Cor will record measurements during the dialysis session, including at least the 15 minutes before and 15 minutes after the session. ZOE (Z0) values will be measured every 6 minutes (± 1 minute) during the dialysis session. ZOE (Z0) values also will be measured every 3 minutes (± 1 minute) before and after the session, for a minimum of 5 measurements. The UFV during the course of hemodialysis will be measured by automated readings provided by the dialysis machine every 6 minutes (± 1 minute). 10. Any IV infusions administered, oral fluid or solid intake, and urine output during the course of hemodialysis will be recorded. Weight, blood pressure, and heart rate will be recorded before and after the dialysis session.The patient's involvement in the study ends after the completion of all procedures planned for the hemodialysis session.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 21 years of age.
* Is currently scheduled to undergo hemodialysis 3 times per week in a clinic setting and has been on this regimen for at least 3 months.
* For those patients with CHF: were diagnosed with CHF by a qualified provider and show symptomatic signs of New York Heart Association (NYHA) Class II to IV at enrollment.
* Is prescribed a net fluid removal of at least 2.5 L during the hemodialysis session.
* Is willing and able to sign informed consent in English.

Exclusion Criteria:

* Is a female patient with a known pregnancy or is unsure of pregnancy status.
* Has known allergies or skin sensitivities to electrode hydrogel and/or acrylic based adhesive.
* Has skin breakdown in areas where device and electrode placement is required.
* Was hospitalized within the 2 weeks prior to enrollment.
* Had intradialytic hypotension requiring administration of intravenous (IV) fluids of ≥250 mL or that resulted in a referral to urgent care, within 2 weeks prior to enrollment.
* Had myocardial infarction, acute coronary syndrome, or stroke within 4 weeks prior to enrollment.
* Has active nephrotic syndrome
* Has severe malnutrition, as diagnosed per a qualified provider.
* Is participating in another clinical trial.
* Has an implanted device that might interfere with the µ-Cor.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhuri Bhat, MS, Study Director — Zoll Medical Corporation
Locations (3):
- United States (3):
  - DaVita Clinical Research, Lakewood, Colorado
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the dialysis clinics of three sites, from November 2016 through February 2017.
Groups:
- Study Arm 1 - Below the Left Axilla: 20 patients undergoing hemodialysis, with at least 10 of these patients having congestive heart failure, will have the u-Cor system placed below the left axilla and the ZOE Fluid Status Monitor
  u-Cor System: Monitoring System
  ZOE Fluid Status Monitor: Monitoring System
- Study Arm 2 - Upper Left Pectoral Area: 20 patients undergoing hemodialysis, with at least 10 of these patients having congestive heart failure, will have the u-Cor system placed on the upper left pectoral area and the ZOE Fluid Status Monitor
  u-Cor System: Monitoring System
  ZOE Fluid Status Monitor: Monitoring System
Period: Overall Study
Arm/Group | Study Arm 1 - Below the Left Axilla | Study Arm 2 - Upper Left Pectoral Area
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm 1 - Below Left Axilla | Study Arm 2 - Upper Left Pectoral Area | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (9.5) | 56 (9.5) | 57 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 15 | 28
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Difference in Correlation of Thoracic Impedance With Ultra-filtration Volume (UFV) Between uCor and ZOE
Description: The primary endpoint measurement is the difference of 1) the Pearson correlation of thoracic impedance made by the u-Cor System to UFV and 2) the Pearson correlation of thoracic impedance made by the ZOE to UFV. Differences in correlation coefficients were calculated for each subject and each study arm.
Time Frame: 15 minutes prior the start of one hemodialysis session to 15 minutes post completion of one hemodialysis session, approximately 2 to 6 hours.
Population: Adult patients undergoing hemodialysis 3x week, with an expected net fluid removal of at least 2.5 L per dialysis session.
Measure: Number (95% Confidence Interval); unit: difference in correlation coefficients
Groups:
- Study Arm 1 - Below Left Axilla: 20 patients undergoing hemodialysis, with at least 10 of these patients having congestive heart failure, will have the u-Cor system placed below the left axilla and the ZOE Fluid Status Monitor
  u-Cor System: Monitoring System
  ZOE Fluid Status Monitor: Monitoring System
Arm/Group | Study Arm 1 - Below Left Axilla | Study Arm 2 - Upper Left Pectoral Area
Number analyzed (Participants) | 20 | 20
difference in correlation coefficients | 0.66 [0.57 to 0.75] | 0.23 [0.12 to 0.35]
Statistical Analysis 1: Comparison: Study Arm 1 - Below Left Axilla; The null hypothesis was that the correlation coefficient of the ZOE device would be greater than the correlation coefficient of the uCor device by at least 0.05. For each subject, a correlation coefficient was calculated between study arm 1 uCor readings and UFV, as well as ZOE readings and UFV. The difference between uCor correlation coefficient and ZOE correlation coefficient for each subject was used as the Primary Measurement; Test type: Non-Inferiority — The µ-Cor System will be considered non-inferior with respect to clinical performance (i.e., trends in fluid change) of the ZOE device if the lower 95% confidence interval of the differences (Primary Measurement) is greater than the non-inferiority margin of -0.05; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.57 to 0.75] — Because the distribution was skewed, the average was calculated by 1) Fisher Transformation of values, 2) averaging the transformed values, 3) back calculating the mean. The Taylor Series expansion and Delta method was used to determine variance
Statistical Analysis 2: Comparison: Study Arm 2 - Upper Left Pectoral Area; The null hypothesis was that the correlation coefficient of the ZOE device would be greater than the correlation coefficient of the uCor device by at least 0.05. For each subject, a correlation coefficient was calculated between study arm 2 uCor readings and UFV, as well as ZOE readings and UFV. The difference between uCor correlation coefficient and ZOE correlation coefficient for each subject was used as the Primary Measurement; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [0.12 to 0.35] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period of 90 days.
Arm/Group | Study Arm 1 - Below Left Axilla | Study Arm 2 - Upper Left Pectoral Area
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03072732/Prot_SAP_000.pdf